CLINICAL TRIAL: NCT05370404
Title: Prescribing Vs. Recommending Over-The-Counter (PROTECT) Analgesics for Patients with Postoperative Pain: a Project on Non-Opioid Pain Medication Use After Discharge from Elective Surgery
Brief Title: Prescribing Vs. Recommending Over-The-Counter (PROTECT) Analgesics for Patients with Postoperative Pain:
Acronym: PROTECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Mark Bicket, MD, PhD, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00203454
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Acute Pain; Surgery
Keywords: Medications after surgery; Surveys; Acetaminophen; NSAIDS; Opioids; Elective outpatient surgery; Magnesium
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prescription Group for acetaminophen, NSAIDs, and magnesium (Active Comparator): Participants will receive prescriptions from the surgical team for non-opioid pain medications to take at home after discharge from surgery.
  The non-opioid pain medications will be acetaminophen 1000 milligram (mg) four times a day (qid) for 3 days then as needed (prn) pain, ibuprofen 600 mg qid for 3 days then prn, and magnesium oxide 400 mg daily prn pain.
  Interventions: Other: Prescription by surgical team
- Over the Counter Group (Active Comparator): Participants will receive a recommendation from the surgical team to take over-the-counter non-opioid pain medications at home after discharge from surgery.
  The non-opioid pain medications will be acetaminophen 1000 mg qid for 3 days then prn pain, ibuprofen 600 mg qid for 3 days then prn, and magnesium oxide 400 mg daily prn pain.
  Interventions: Other: Recommendation by surgical team

INTERVENTIONS:
Other: Prescription by surgical team — The surgical team prescribes medications to the patient
  Arms: Prescription Group for acetaminophen, NSAIDs, and magnesium
Other: Recommendation by surgical team — The surgical team recommends the patient to take over-the-counter medications
  Arms: Over the Counter Group

SUMMARY:
This is a research project in which two standard of care practices will be evaluated to examine the difference in outcomes. The goal is to improve patient care and safety. One group will receive prescriptions for acetaminophen, nonsteroidal anti-inflammatory drugs (NSAIDs), and magnesium. The other group will receive the recommendation to take acetaminophen, NSAIDs, and magnesium as over-the-counter drugs in the same dosage as the prescription group. The same doses and routes for non-opioid medications will be used in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Anticipated to be prescribed and use an opioid medication to treat acute pain after elective outpatient surgery

Exclusion Criteria:

* Contraindications to taking acetaminophen or NSAIDs
* Significant analgesic medication use before surgery
* Inability to receive emails or phone calls for follow up assessment
* Patients who have reoperation, another surgery, or experience complications within 14 days after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Maximal consumption of acetaminophen and NSAIDs within 3 days after discharge from surgery | 3 days following surgery discharge
  Patient report of the number of doses within the first 3 days of the use of both acetaminophen and NSAID at home after discharge from surgery. Patients are anticipated to take up to 4 doses of acetaminophen and NSAIDs per day. Over 3 days, patients would be anticipated to take a maximum of 12 doses. This outcome is a count that ranges from 0 (no doses of acetaminophen plus NSAIDs) to 12.
Patient use of acetaminophen within 3 days after discharge from surgery | 3 days following surgery discharge
  Patient-reported use of acetaminophen at any point in time within the first 3 days at home after discharge from surgery.
Patient use of NSAIDS within 3 days after discharge from surgery | 3 days following surgery discharge
  Patient-reported use of NSAIDs at any point in time within the first 3 days at home after discharge from surgery.
Patient use of acetaminophen and NSAID with opioid within 3 days after discharge from surgery | 3 days following surgery discharge
  Patient-reported use of both acetaminophen and NSAID on every day oral pain medication is taken within the first 3 days at home after discharge from surgery.
Delayed acetaminophen and NSAID use as reported at 12-16 days after discharge from surgery | 12-16 days following surgery discharge
  Patient-reported use of acetaminophen and/or NSAIDs in the second week after discharge from surgery.

SECONDARY OUTCOMES:
Patient-reported consumption of opioid pills within 3 days after discharge from surgery | 3 days following surgery discharge
  The total amount of opioids consumed over days 0-3 after discharge from surgery will be compared between the two groups.
Patient-reported consumption of opioid pills as reported at 12-16 days after discharge from surgery | 12-16 days following surgery discharge
  The total amount of opioids consumed over the second week after discharge from surgery will be compared between the two groups.
Pain intensity at site of surgery 3 days following surgery discharge | 3 days following surgery discharge
  This is a one question survey in which the participants are asked to rate the pain at the site of the surgery that best describes the pain from a scale of 0 (no pain) to 10 (pain is the worst). Trends in worst pain intensity over days 0-3 after discharge from surgery will be compared between the two groups.
Pain intensity at site of surgery as reported at 12-16 days following surgery discharge | 3 days following surgery discharge
  This is a one question survey in which the participants are asked to rate the pain at the site of the surgery that best describes the pain from a scale of 0 (no pain) to 10 (pain is the worst). Trends in worst pain intensity over the second week after discharge from surgery will be compared between the two groups.
Medication side effects within 3 days following surgery discharge | 3 days following surgery discharge
  Patient report of common analgesic related side effects will be measured using the Medicare symptom checklist. Composite report of any side effect over days 0-3 after discharge from surgery will be compared between the two groups.
Patient satisfaction with pain treatment within 3 days following surgery discharge | 3 days following surgery discharge
  This is a one question survey in which the participants are asked to rate the satisfaction for pain management with a scale from very dissatisfied to very satisfied. Patient report of overall satisfaction with the postoperative pain treatment over days 0-3 after discharge from surgery will be compared between the two groups.
Patient use of magnesium within 3 days after discharge from surgery | 3 days following surgery discharge
  Patient-reported use of magnesium at any point in time within the first 3 days at home after discharge from surgery.
Delayed magnesium use days as reported at 12-16 days after discharge from surgery | 12-16 days following surgery discharge
  Patient-reported use of magnesium in the second week after discharge from surgery.

OTHER OUTCOMES:
Opioid disposal | 3-16 days following surgery discharge
  Patient-reported disposal of opioids after completion of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bicket, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No